CLINICAL TRIAL: NCT06826131
Title: Determination of the Optimal Cut Off Value of the Modified Ashworth Scale in the Evaluation of Gait Performance and Functional Mobility in Individuals With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Betul Ergun, research assistant, Inonu University
Other Study IDs: Ashworth- SP
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy (CP); Walking Performance; Functional Mobility
Keywords: cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Participants' biospecimens and DNA will not be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cerebral Palsy: Individuals with Cerebral Palsy between the ages of 6-15 with gMFSS:1-2

SUMMARY:
The spastic type, which is the most common type of CP, constitutes approximately 75% of individuals. The most prominent physical examination finding in patients with CP is marked tonus changes. Increased tonus and involuntary movement patterns are frequently observed clinically. Today, the Modified Ashworth Scale is mostly used in the evaluation of spasticity in individuals. Ashworth scale was defined in 1964 and modified in 1987. This scale was developed to assess muscle tone. Resistance to passive movement is evaluated and scored between 0-4.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is one of the common causes of disability in childhood. The prevalence of the disease has been evaluated as 2-3 per 1000 live births on average in various societies. In various prevalence studies conducted in our country, the prevalence of the disease was found to be 1.1- 4.4 per 1000 live births.

CP is a disease with multifactorial etiology. Although antenatal, perinatal and neonatal effects often play a role together, the most important known risk factors are low birth weight and prematurity. Intrauterine infections have been identified as the most important cause of CP etiology in individuals with prematurity and low birth weight. These infections can trigger premature birth and cause damage to the central nervous system, which has not yet completed its development.

In CP, classifications are made according to the extremity involvement, clinical features, etiologies and many different pathogenesis. Currently, the most common and widely used classification is the one defined by Phelps and Perlstein according to the involved extremity and tonus disorder.

A) Spastic type: (pyramidal): Monoplegia, Diplegia, Hemiplegia, Triplegia, Tetraplegia B) Dyskinetic type: (Extrapyramidal): Athetoid, Choreic, Choreoathetoid, Dystonic C) Ataxic type D) Hypotonic type E) Mixed type Materials and Methods The study was designed to determine the optimal cut off value of the modified ashworth scale in the evaluation of gait performance and functional mobility in individuals with CP aged 6-15 years. Patients admitted to the CP outpatient clinic of Kayseri City Hospital, Physical Medicine and Rehabilitation Clinic and Twenty-five individuals who meet the inclusion criteria will be included in the study.

Modified Ashworth Scale 0 : Normal muscle tone. 1 : Slight increase in muscle tone, minimal resistance is felt at the end of joint movement.

1+ : Minimal resistance in less than half of the joint movement. 2 : Significant increased muscle tone throughout the entire movement, but the joint can still be moved easily.

3 : There is significant increased muscle tone throughout the entire movement making passive movement difficult.

4 : The affected muscles are completely rigid, remaining in fixed flexion or extension.

Gross Motor Function Measure Classification System (GMFCS) KMFSS, which is one of the most widely used scales to classify the severity of movement disorders in individuals with CP and to evaluate the current activity levels of the subjects, was developed by Palisano et al. in 1997. In 2012, El et al. conducted a validity and reliability study of the CMFCS for the Turkish population.

Gross motor function classification system Level 1 Walks independently. There is limitation in advanced gross motor skills.

Level 2 Walks without an assistive device. Has limitations when walking in public.

Level 3 Walks with an assistive device. There is limitation while walking in the community.

Level 4 Has limitations. Self-mobile. Transported in the community or uses a wheelchair.

Level 5 Mobilization is severely limited even with assistive technologies. 10 meter walk test: It is used to measure walking speed from functional parameters. A 16-meter walking track is created to perform the test. The first 3 and last 3 meters of this track are completed without taking into account and the measurements are repeated 3 times each. Before the test is performed, starting and ending points are determined on non-slippery ground. The individual starts walking, the stopwatch is started after the first three meters. The stopwatch is stopped at the end of the tenth meter. After the individual walks the last 3 meters, walking is terminated. The completion time of the test is recorded in seconds.

Assessment of Mobility TUG test: It was performed using a standard chair (46 cm high). Patients sat with their backs against the chair. Patients were instructed to get up from the chair without support, walk three meters marked on the floor, turn around, walk back to the chair and sit down again. Patients were told that the test should be performed at a normal pace. The stopwatch was started with the word "start" and stopped when the patient sat down. TUG time was measured in seconds (s).

Five Times Sit and Stand Test: It is used for functional mobility measurements. In the test, the individual sits with arms crossed over the shoulders and back leaning against the chair. With the "go" command, the patient stands up and sits down five times quickly from the standard chair. The elapsed time is measured with a stopwatch.

ELIGIBILITY:
Inclusion Criteria:

* GMFSS:1-2,
* Have the appropriate cognitive level to adapt to the tests to be performed in the study,
* Individuals between the ages of 6-15 who agreed to participate in the study were included.

Exclusion Criteria:

* Bone and/or soft tissue surgery on the lower extremities within the last 1 year who had the operation,
* Extensive serious skin injuries, skin infection,
* Lower extremity MAS score > 2,
* Mental retardation,
* Individuals who had botulinum toxin applied to their lower extremities within the last 1 year were excluded.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: It was observed that the effect size obtained in the reference study was strong (d=1.28). As a result of the power analysis performed considering that an effect size at this level could also be obtained; it was calculated that 95% power could be obtained at 95% confidence level when at least 25 people were included in the study (Freire et al, 2023).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Optimal cut off value of modified ashworth scale in individuals with CP | 1 days
  To determine the optimal cut off value of the modified ashworth scale in the evaluation of gait performance and functional mobility in individuals with CP aged 6-15 years. The Modified Ashworth Scale is a 6-point scale. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity or increased resistance to passive movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Physical Medicine and Rehabilitation Clinic, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided